CLINICAL TRIAL: NCT00452192
Title: Detailed Analysis of the Effects of Telmisartan on Renal Perfusion in Patients With Metabolic Syndrome
Brief Title: Telmisartan and Renal Perfusion in Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SFB 423-TP B5 Niere MRT
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Telmisartan — telmisartan 80 mg daily over 2 weeks

SUMMARY:
A major complication of diabetes mellitus is diabetic nephropathy. In previous studies the investigators could demonstrate that in patients with type 2 diabetes mellitus despite unaltered basal and stimulated nitric oxide (NO) - activity, the renal response to the antioxidant vitamin C was more pronounced compared to control subjects. These data suggest that oxidative stress is increased in the renal vasculature of diabetic patients. Furthermore, NO-activity in diabetic patients appears to be up regulated to compensate for increase in oxidative stress. This hypothesis is supported by the demonstration of increased endothelial nitric oxide synthase (eNOS) expression in kidney biopsies of diabetic patients.

Angiotensin receptor blockers have been found to reduce oxidative stress in various vascular beds. Some drugs of this class, Telmisartan for example, also exhibit partial agonist properties to the PPARγ receptor and might be of great benefit for patients with diabetes mellitus or metabolic syndrome due to an additional improvement in insulin resistance. Despite its effect on oxidative stress angiotensin receptor blockers beneficially alter renal haemodynamics by reducing intraglomerular pressure and thus protect against glomerular injury.

Recent advances in magnetic resonance imaging lead to the development of new techniques that allow a separate measurement of renal medullar and cortical perfusion. This magnetic resonance imaging technique might be a useful tool to detect alterations at an early level in the kidneys of patients at high risk for diabetic nephropathy. In the current study, the investigators want to evaluate the new magnetic resonance imaging technique by measuring medullar and cortical renal perfusion before and after pharmacological intervention with telmisartan in patients with metabolic syndrome.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

1. Male subject of 18 to 65 years of age
2. Subjects with at least 3 of 5 criteria of the metabolic syndrome:

   * Central (abdominal) obesity: waist circumference >= 102 cm
   * Hypertension: >=135/>=85 mmHg
   * Hypertriglyceridemia: >= 150 mg/dL
   * Low HDL -cholesterol: < 40 mg/dL
   * Hyperglycemia: fasting glucose >= 110 mg/dL and
3. Subjects with a history of essential hypertension or newly diagnosed with essential hypertension with a BP reaching following criteria:

   * MSSBP >=135 mmHg and < 180 mmHg and/or MSDBP >= 85 mmHg and < 110 mmHg
4. Subjects who are eligible, able to participate in the study, and who consent to do so after the purpose and nature of the investigation has been clearly explained to them. Existence of written informed consent.
5. Subjects with normal renal function (according to the MDRD IV eGFR > 60 ml/min/1.73m^2)

Exclusion Criteria:

1. Subjects treated with an ACE or an ARB within 3 month of study entry who are unable or unwilling to undergo the 3 month washout period.
2. Known secondary hypertension of any etiology (e.g., uncorrected renal artery stenosis).
3. Any of the following conditions: Atrial fibrillation, AV block II or higher, history of myocardial infarction, instable angina pectoris, pathologic ECG changes, heart failure NYHA III/IV
4. Severe Depression
5. History of epileptic seizures
6. Proliferative Retinopathy
7. MSSBP pressure > 180 mmHg or MSDBP > 110 mmHg
8. Known Renal arterial stenoses (on one or both sides)
9. Known or suspected contraindications or intolerance to or history of hypersensitivity to any of the study drugs or to drugs belonging to the same therapeutic class (e.g., ARBs) as the study drug.
10. Subjects who take drugs that are not approved/admitted in germany or subjects participating now or three month prior to this trial in other studies.
11. Therapy with not allowed concomitant drugs.
12. Current abuse or recent history of alcohol or other drug substance abuse (past 12 month).
13. Subjects that in the eye of the investigation seem to be noncompliant and unwilling or not able to show up for control examinations. Subjects with a history of non-compliance to medical regimes or unwillingness to comply with the study protocol.
14. Subjects whose body structure (e.g., weight, height, body circumference, etc.) exceeds the restrictions of the local site of MRI instrument.
15. Use of pacemakers, ICD, defibrillators, or any device which interferes with an MRI. Subjects that have any metallic material anywhere in their body that might interfere with an MRI.
16. Significant claustrophobia.
17. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs including, but not limited to, any of the following:

    * History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection.
    * Currently active or previously active inflammatory bowel disease during the 12 months prior to study entry.
    * Currently active gastritis, duodenal or gastric ulcers, or gastrointestinal/rectal bleeding during the 3 months prior to study entry.
    * Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase.
    * Evidence of hepatic disease as determined by any one of the following:

      * SGOT
      * or GPT values exceeding > 150 % of the upper limit of the normal range GGT
      * or AP or bilirubin levels exceeding 200 % of the upper limit of the normal range.
    * Evidence of renal impairment as determined by anyone of the following:

      * serum creatinine > 1.7 mg/dl for males and serum creatinine of > 1.5 mg/dl for females at study entry
      * a history of dialysis, or
      * a history of nephritic syndrome.
    * Current treatment with cholestyramine and colestipol resins.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in RPF to L-NMMA at baseline and after telmisartan (MRI) | 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Roland. E Schmieder, MD, Principal Investigator — Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nürnberg
Locations (1):
- Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nürnberg, Erlangen, Germany

REFERENCES:
- See also: Related Info — http://www.crc-erlangen.de